CLINICAL TRIAL: NCT03486379
Title: FOLFIRI as a Second-line Therapy in Patients With Docetaxel-pretreated Gastric Cancer
Brief Title: Folfiri as Third Line of Treatment
Status: Completed | Type: Observational
Sponsor: IRCCS Cancer Referral Center of Basilicata (Other)
Responsible Party: Principal Investigator, Giandomenico Roviello, MS, PhD, IRCCS Cancer Referral Center of Basilicata
Other Study IDs: IRCCS-CROB
Record Dates: First submitted 2018-03-23; First posted 2018-04-03 (Actual); Last update posted 2018-04-03 (Actual); Status verified 2018-03

CONDITIONS: Gastric Cancer; Ramucirumab; Third Line
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to investigate the activity of Folfiri as Third line of treatment in mGC progressed after ramuciramb-based second line.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed, ramucirumab pretreated metastatic gastric cancer who received
* Eastern Cooperative Oncology Group performance status ≤2 (ECOG PS)
* aged > 18 years
* neutrophil count ≥1500/μl
* platelet count ≥100 000/μl),
* renal (serum creatinine ≤1.5 mg/dl)
* liver (serum bilirubin ≤2 mg/dL) functions
* normal cardiac function,
* absence of second primary tumor other than non-melanoma skin cancer
* no concurrent uncontrolled medical illness.

Exclusion Criteria:

* Eastern Cooperative Oncology Group performance status >2 (ECOG PS)
* No prior treatment with ramucirumab
* operable metastatic disease were excluded from the study
* severe cardiac dysfunction, congestive heart failure or a recent myocardial infarction
* uncontrolled sites of infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with metastatic gastric cancer progressed after two lines of treatment including ramucirumab-based therapy.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2016-03; Primary Completion 2017-09-30 (Actual); Study Completion 2018-03-23 (Actual)

PRIMARY OUTCOMES:
response rate (confirmed complete and partial response). | From date of enrollment to best radiological evaluation, up to 12 months
  rate of patients with complete or partial response

SECONDARY OUTCOMES:
Progression free survival | From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months
  Time from start of treatment to Progression or death
Overall survival | From date of enrollment until the date of death from any cause, whichever came first, assessed up to 12 months
  Time from start of treatment to Death for any cause
Toxicity | From date to start therapy up to 12 months
  Incidence of Toxicity according National Cancer Institute Common Terminology Criteria